CLINICAL TRIAL: NCT00419445
Title: A Double-Blind, Randomized, Proof-of-Concept Crossover Trial to Assess the Effects of GTS21 on Cognitive Function, Clinical Symptoms, and Adverse Events in Adults Diagnosed With Attention-Deficit Hyperactivity Disorder
Brief Title: Safety and Efficacy of GTS21 in Adults With Attention-deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CoMentis (Industry)
Responsible Party: Carl Grove, CoMentis (formerly Athenagen)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GTS21-202
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Results first posted 2010-09-10 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder in adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GTS21 25 mg tid/Placebo 25 mg tid (Active Comparator)
  Interventions: Drug: GTS21/Placebo
- GTS21 75 mg tid/Placebo 75 mg tid (Active Comparator)
  Interventions: Drug: GTS21/Placebo
- GTS21 150 mg tid/Placebo 150 mg tid (Active Comparator)
  Interventions: Drug: GTS21/Placebo

INTERVENTIONS:
Drug: GTS21/Placebo

SUMMARY:
This study will be a randomized, double-blind, placebo-controlled crossover study to assess the effects of GTS21 (25 mg three times a day (tid), 75 mg tid, 150 mg tid) compared to placebo in non-smoking adults aged 18-55 with a diagnosis of ADHD, any subtype.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18-55, inclusive.
* Diagnostic and Statistical Manual for the Classification of Mental Disorders, Fourth Edition (DSM-IV) criteria for ADHD, any subtype, based on a detailed psychiatric evaluation including the Conners' Adult ADHD Interview for DSM-IV (CAADID) and the Structured Clinical Interview for DSM-IV (SCID).
* A minimum Total ADHD Symptoms Index score of 28 on the clinician administered CAARS.
* A Clinical Global Impressions-Severity (CGI-S) score of ≥ 4 at Screening.
* Normal or clinically insignificant ECG and clinical laboratory (e.g., liver enzymes, complete blood count, etc.) findings at Screening.
* Intellectual function at age-appropriate levels, as deemed by the Investigator.
* Supine systolic and diastolic blood pressure measurements < 140 and < 90, respectively, at Screening.
* Written, signed and dated informed consent for the patient to participate in the study must have been given by the patient.
* Females of child-bearing potential must have had a negative serum beta human chorionic gonadotropin (HCG) pregnancy test at Screening and be practicing double-barrier methods of contraception, if sexually active and for 30 days following administration of any study drug.
* Male patients who were sexually active must have agreed to use a reliable form of contraception during the study and for 30 days following administration of any study drug.
* Be fluent in English (speaking, writing and reading).

Exclusion Criteria:

* Any current, controlled (requiring a prohibited medication) or uncontrolled, comorbid psychiatric diagnosis (except simple phobias), all major depressive disorders [dysthymia and mood disorder not otherwise specified (NOS) allowed unless medication required],and any severe comorbid Axis II disorders or severe Axis I disorders such as Post Traumatic Stress Disorder, bipolar illness, psychosis, obsessive-compulsive disorder, substance abuse disorder, or other symptomatic manifestations that, in the opinion of the Investigator, contraindicated treatment with GTS21 or confound efficacy or safety assessments.
* Any condition or illness (including clinically significant abnormal laboratory values) which, in the opinion of the Investigator, represented an inappropriate risk to the patient and/or could confound the interpretation of the study.
* Regular use of nicotine products (including 90 days before Screening), including smoking, transdermal patch, chewing tobacco, etc. (verified via salivary cotinine levels at Screening).
* Current use of any prohibited medication or other medications, including herbal supplements, that have central nervous system (CNS) effects or affect cognitive performance, such as sedating antihistamines and decongestant sympathomimetics (bronchodilators were permitted).
* Use of another investigational product or participation in a clinical study within 30 days prior to Screening.
* Body Mass Index (BMI) > 32.
* Known or suspected allergy, hypersensitivity, or clinically significant intolerance to nicotine or nicotinic agonists.
* Clinically important abnormality on urine drug screen (excluding the patient's current ADHD stimulant, if applicable) at Screening.
* Pregnant or currently lactating.
* Patients that had previously been enrolled into this study and subsequently withdrawn.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Grove, Study Director — CoMentis (formerly Athenagen)
Locations (2):
- United States (2):
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- See also: Related Info — http://www.comentis.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 25 mg Tid | 75 mg Tid | 150 mg Tid
Started | 8 | 16 | 8
Completed | 7 | 14 | 7
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg Tid | 75 mg Tid | 150 mg Tid | Total
Number analyzed (Participants) | 8 | 16 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 16 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.5 (9.47) | 371. (10.24) | 34.8 (15.42) | 39.2 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 3 | 12
  Male | 6 | 9 | 5 | 20
Region of Enrollment [Number; unit: participants]
  United States | 8 | 16 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Safety and Tolerability of GTS21 (25 mg Tid, 75 mg Tid, 150 mg Tid).
Description: The proportion of subjects with Treatment Emergent Adverse Events.
Time Frame: Baseline to study completion
Measure: Number; unit: % of subjects
Arm/Group | 25 mg Tid | 75 mg Tid | 150 mg Tid
Number analyzed (Participants) | 8 | 16 | 8
% of subjects | 67 | 72 | 100

ADVERSE EVENTS:
Arm/Group | 25 mg Tid | 75 mg Tid | 150 mg Tid
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 13/18 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg Tid (N=8) | 75 mg Tid (N=18) | 150 mg Tid (N=8)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days